CLINICAL TRIAL: NCT06013072
Title: The Effects of 3-month Supplementation With a Pre-probiotic on Patient- and Clinician-reported Outcomes, and Brain Tissue Metabolism in Patients With Post-covid Fatigue Syndrome: a Placebo-controlled Randomized Clinical Trial
Brief Title: Pre-probiotic Supplementation for Post-covid Fatigue Syndrome
Acronym: STOPPFATIQUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Principal Investigator, Sergej Ostojic, Professor, University of Novi Sad, Faculty of Sport and Physical Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2022-03-23_CFS
Record Dates: First submitted 2023-08-25; First posted 2023-08-28 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Long COVID
Keywords: Prebiotic; Probiotic; Metabolism; Fatigue
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-probiotic (Experimental): One sachet per day during breakfast
  Interventions: Dietary Supplement: Dietary Supplement: Experimental
- Placebo (Placebo Comparator): One sachet per day during breakfast
  Interventions: Dietary Supplement: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Experimental — Combination of pre-probiotic
  Arms: Pre-probiotic
Dietary Supplement: Dietary Supplement: Placebo — Inert compound
  Arms: Placebo

SUMMARY:
The goal of this randomized controlled double-blind parallel-group interventional trial is to evaluate the effects of of dietary supplementation with a pre-probiotic on patient- and clinician-reported outcomes, and brain tissue metabolism in patients with post-covid fatigue syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years
* Covid-19 positive test within last 3 months (as documented byvalid PCR or antigentest
* Moderate-to-severe fatigue (20-MFI test total score > 43.5)
* At least one of additional covid-19 related symptoms (anosmia,ageusia,breathingdifficulties,lungpain, body aches, headaches, difficulties concentrating etc.)

Exclusion Criteria:

* Other pulmonary and cardiovascular conditions
* History of dietary supplement use during the past 4 weeks
* Organic gastrointestinal (GI) disorders such as inflammatory bowel disease, coeliac disease, eosinophilic disorders, or current infection of the GI tract.
* Bowel surgery or short bowel syndrome.
* Medication or supplement which can impact the gut microbiome, including: antibiotics, antimicrobials, or antifungals in the two months
* Probiotic or prebiotic supplements in the last 4 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Fatigue | Change from baseline fatigue at 3 months
  Level of fatigue as assessed by the Multidimensional Fatigue Inventory (MFI)

SECONDARY OUTCOMES:
Brain creatine | Change from baseline brain creatine concentrations at 3 months
  Magnetic resonance spectra for brain creatine concentrations
Patient-reported symptoms | Change from baseline fatigue at 3 months
  Scale of symptoms assessed by Visal Analog Scales (VAS), minimum 0 maximum 10; higher scores mean a worse outcome
Time to exhaustion | Change from baseline time to exhaustion at 3 months
  Running time to exhaustion during incrementaltestontreadmill

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Bioenergetics Lab at Faculty of Sport and PE, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in long COVID. Data will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.

REFERENCES:
- [Derived] Ranisavljev M, Stajer V, Todorovic N, Ostojic J, Cvejic JH, Steinert RE, Ostojic SM. The effects of 3-month supplementation with synbiotic on patient-reported outcomes, exercise tolerance, and brain and muscle metabolism in adult patients with post-COVID-19 chronic fatigue syndrome (STOP-FATIGUE): a randomized Placebo-controlled clinical trial. Eur J Nutr. 2024 Nov 26;64(1):28. doi: 10.1007/s00394-024-03546-0. PMID 39592468